CLINICAL TRIAL: NCT00520208
Title: A Phase II Study of Oral Tamibarotene in Acute Promyelocytic Leukemia Patients Who Have Received Prior Therapy With ATRA and Arsenic Trioxide (STAR-1)
Brief Title: Safety, Efficacy, & Pharmacokinetic Study of Tamibarotene to Treat Patients With Relapsed or Refractory APL
Acronym: STAR-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytRx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNO-507-P2
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: ATRA; Trisenox; Arsenic; Arsenic Trioxide; APL
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — tamibarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tamibarotene — For induction therapy, tamibarotene will be self-administered via tablets on an outpatient basis at a dose of 6 mg/m2 per day, taken orally, in two divided doses approximately one hour after breakfast and dinner. Induction therapy will continue for a maximum of 56 days until either a morphologic leukemia-free state or complete response (CR) has been achieved. For patients who achieve a CR with induction therapy, consolidation therapy will commence 4 to 8 weeks after the end of induction therapy. For patients who have a morphologic leukemia-free state after induction therapy but who fail to achieve a CR, consolidation therapy will commence 8 weeks after the end of induction therapy.
  Other Names: Amnolake

SUMMARY:
This is a Phase II, open-label, non-randomized study to evaluate the safety, efficacy, and pharmacokinetics of tamibarotene in adult patients with relapsed or refractory acute promyelocytic leukemia (APL) following treatment with all-trans-retinoic acid (ATRA) and arsenic trioxide (ATO). Patients must have received and failed therapy with ATRA and ATO. Treatment may have been administered either as combination therapy or sequentially as single agents. Patients who are intolerant to either drug are eligible for this study.

ELIGIBILITY:
Patients must meet all of the following criteria for admission into the study:

1. Have a diagnosis of either relapsed and/or refractory APL:

   * Refractory disease is defined as a confirmed diagnosis of APL and a myeloblast plus promyelocyte count of > 10% in the bone marrow in patients who have failed to respond to induction therapy in the first or second line setting. Induction therapy must have included ATRA- and ATO-based therapy given either sequentially or in combination.
   * Relapsed disease is defined as a confirmed diagnosis of APL and a myeloblast plus promyelocyte count of > 10% in the bone marrow following a documented complete remission or positive RT-PCR assay for PML/RAR-α in two consecutive tests separated by at least one month, after treatment with ATRA- and ATO-based therapy given either sequentially or in combination.
2. Confirmation of diagnosis and relapsed/refractory APL must be obtained in blood or bone marrow mononuclear cells by at least one of the following methods:

   * Conventional cytogenetics showing the translocation t(15:17),
   * Positive RT-PCR assay for PML/RAR-α, or
   * Fluorescence in situ hybridization (FISH) analysis showing evidence of the PML/RAR-α translocation.
3. Patients must have received and failed therapy with ATRA and ATO either within the same or separate induction/consolidation schedule(s). Treatment must have been administered for a minimum of 28 days for each agent. Treatment may have been administered either as combination therapy or sequentially as single agents. Patients who failed to complete a course of induction/consolidation therapy, as specified, due to drug intolerance are eligible for the study.
4. Patients in whom ATO is contraindicated (for example due to congenital long QT syndrome) are eligible for inclusion on study if they have received and failed ATRA therapy as defined in (3).
5. Be able to provide written informed consent prior to enrollment into the study.
6. Be ≥ 18 years old.
7. Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
8. Have an estimated life expectancy of ≥ 12 weeks.
9. Be male or a non-pregnant, non-lactating female. Fertile patients must agree to use an effective barrier method of contraception (e.g., latex condom, diaphragm, or cervical cap) to avoid pregnancy while on therapy and for 90 days following the discontinuation of the study drug. [In countries where double barrier contraception is required by Regulatory Authorities, patients who are fertile must agree to use 2 forms of barrier method contraception (e.g., latex condom AND a diaphragm or cervical cap) while on therapy and for 90 days following the discontinuation of the study drug.]

   A non-fertile female is defined as:
   * Postmenopausal (amenorrheic for ≥ 12 months)
   * Undergone a complete oophorectomy or hysterectomy.
10. Have a negative serum or urine pregnancy test within 10 days prior to the first dose of study drug (if patient is a female of childbearing potential).
11. Have adequate organ function.

Patients who meet any of the following criteria will be excluded from study admission:

1. Extramedullary leukemia.
2. Patients on a vitamin A preparation or patients with hypervitaminosis A.
3. Have received cytotoxic therapy ≤ 2 weeks from the start of therapy. If the patient needs these agents due to urgent medical care within 2 weeks prior to starting tamibarotene, a waiver may be granted by the INNOVIVE Medical Monitor.
4. Have a history of myelodysplastic syndromes (MDS).
5. Have impaired cardiac function or clinically significant heart disease including:

   * Myocardial infarction within 3 months, unstable angina pectoris, congenital long QT syndrome and clinically significant resting bradycardia (< 50 beats per minute), uncontrolled congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with antihypertensive medication.
6. Have an active, uncontrolled systemic infection considered opportunistic, life-threatening, or clinically significant at the time of treatment.
7. Have clinically significant acute or chronic liver or renal disease considered unrelated to leukemia.
8. Have uncontrolled hyperlipidemia.
9. Have uncontrolled or poorly controlled diabetes mellitus.
10. Have impaired gastrointestinal function that may significantly alter drug absorption (e.g., uncontrolled vomiting, ulcerative colitis, malabsorption, or small bowel resection).
11. Are pregnant or lactating.
12. Have psychiatric disorder(s) that would interfere with consent, study participation, or follow-up.
13. Have not recovered from acute toxicities of all previous therapy prior to enrollment.
14. Have any other severe concurrent disease and/or uncontrolled medical conditions, which, in the judgment of the investigator, could predispose patients to unacceptable safety risks or compromise compliance with the protocol.
15. Have a history of another primary malignancy that has been actively treated in the last 24 months.
16. Are unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-09; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To determine the rate of durable complete response for tamibarotene therapy when administered as a single agent to adult patients with relapsed or refractory APL. | Minimum 28 days

SECONDARY OUTCOMES:
(1) To determine the rates of morphologic leukemia-free state, partial response, cytogenetic complete response, and molecular complete response for tamibarotene therapy in the indicated patient population. | Minimum 28 days
(2) To determine the safety profile and tolerability of tamibarotene in the indicated patient population. | Up to 32 weeks
(3) To determine the pharmacokinetic (PK) profile of tamibarotene when administered in the indicated patient population. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - UT MD Anderson Cancer Center, Houston, Texas